CLINICAL TRIAL: NCT04565067
Title: Identification and Characterization of SARS-CoV-2 Specific CD8 T Cells in Humans a Clinical Observation Trial
Brief Title: Identification and Characterization of SARS-CoV-2 Specific CD8 T Cells in Humans
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000140; 000140-AG
Record Dates: First submitted 2020-09-24; First posted 2020-09-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11-17

CONDITIONS: COVID-19
Keywords: CD8 T Cell; COVID-19; Immune Response; Epitope; Aging; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: COVID-19 recovered adult patients

SUMMARY:
Background:

The higher death rate from COVID-19 in the older population is associated with low CD8 T cell counts in the blood. Researchers want to learn the status of CD8 T cells specific to SARS-CoV-2 and their changes with aging and in COVID-19. This may help to identify why COVID-19 is particularly lethal in the elderly and help to create an effective vaccine against SARS-CoV-2 in the elderly.

Objective:

To identify SARS-CoV-2 specific CD8 T cells in humans, and to determine their quantity and quality in people who have recovered from COVID-19.

Eligibility:

Maryland residents age 18 and older who have tested positive for and recovered from COVID-19.

Design:

Participants will be screened by phone. They must be able to provide a copy of their positive COVID-19 test result.

Participants will visit the NIA/Clinical Research Unit. The visit will take about 1 hour.

Laboratory tests showing a positive COVID-19 result will be verified.

Participants vital signs will be checked. This will include blood pressure, temperature, pulse, and respiration. Height and weight will be measured.

Participants will have a medical history and medicine review. They will complete a COVID-19 questionnaire.

Participants will have blood drawn. They will give a urine sample.

Participants will give a saliva sample. They will rinse their mouth with water. After about 3 minutes, they will let saliva pool in the base of their mouth and then spit into a sterile container.

Participants may be asked if they would be willing to return for optional visits at about 4 months and 1 year later. They will repeat the same laboratory sampling performed at the first visit.

...

DETAILED DESCRIPTION:
Study Description:

This study is to identify epitopes of SARS-CoV-2 that are recognized by CD8 T cells in the blood of healthy young and old participants as well as COVID-19 recovered. We will also measure general health factors using blood, saliva and urine samples. By analyzing the frequency, differentiation, and expansion of these SARS-CoV-2 recognizing CD8 T cells, we hope to shed light into the T cell immunity against SARS-CoV-2 and its change with age and post-infection.

Objective:

To identify SARS-CoV-2 specific CD8 T cells in humans, and to determine their quantity and quality in recovered COVID-19 patients.

Endpoints:

Primary Endpoint: We are investigating the presence or absence of various SARS-CoV-2 specific CD8 T cells in healthy adults and in COVID-19 recovered patients to understand the composition of CD8 T cell immunity in COVID-19 pathogenesis. We plan to determine CD8 T cells that are responsive to SARS-CoV-2.

Secondary Endpoint: To determine the number and quality of SARSCoV-2 specific CD8

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability of subject to understand the study and stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female, aged 18 years or older.
3. Able to speak and read English.
4. Willingness and ability to come to the NIA Clinical Research Unit at MedStar Harbor Hospital in Baltimore for study procedures.
5. Proof of positive SARS-CoV-2 testing exhibiting no current clinical symptoms.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unable to verify identification of volunteer by state issued ID card, driver's license, or military ID. Participants earning greater than $600.00/year are issued a 1099 form, therefore, positive identification is required.
2. Unable to provide informed consent
3. Current use of steroids, immunosuppressive medications, radiation therapy, or chemotherapy medications.
4. Pregnancy.
5. Received immunization therapy for COVID-19 or have received a COVID-19 vaccination prior to Visit 1.

In addition, eligible participants may not be immediately able to participate in the study but might be eligible at a later date. These include:

1. Symptoms of a viral infection on visit 1 (defer until resolved).
2. Medication: Volunteers taking the following medications would be deferred for 2 weeks after course has been completed and volunteer is feeling well: Antibiotics, antifungals, antimalarials, antvirals.
3. Temporary steroids (tapers): Deferred for 72 hours after symptoms are resolved and prescription is completed if taken orally, intravenously, or intramuscular. No deferral if taken intranasal, inhaled, or for joint injection.
4. Infection or Fever: Deferred until 2 weeks after antibiotics are completed and /or volunteer is feeling well.
5. We wish to only select recovered confirmed COVID-19 patients. Therefore, those who may have a household member (co-habitant) who is newly diagnosed with COVID-19 or who has symptoms will be deferred for 14 days.
6. Treatment with another investigational drug or other intervention within 14 days of visit 1 per the discretion of the Principal Investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 recovered adult patients: sample size =100, both genders, 18 years of age and older, all races, and residents of the state of Maryland.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Determine CD8 T cells that are responsive to SARS-CoV-2. | 4 month and 1 year data
  We are investigating the presence or absence of various SARS-CoV-2 specific CD8 T cells in healthy adults and in COVID-19 recovered patients to understand the composition of CD8 T cell immunity in COVID-19 pathogenesis.

SECONDARY OUTCOMES:
Determine CD8 T cells that are responsive to SARS-CoV-2. | Ongoing
  To determine the number and quality of SARS-CoV-2 specific CD8 T cells in relationship with the severity of COVID-19 disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nan-Ping P Weng, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
NIA IRP are in discussion and a plan has not been finalized.

REFERENCES:
- [Derived] Yao Q, Doyle ME, Liu QR, Appleton A, O'Connell JF, Weng NP, Egan JM. Long-Term Dysfunction of Taste Papillae in SARS-CoV-2. NEJM Evid. 2023 Sep;2(9):10.1056/evidoa2300046. doi: 10.1056/evidoa2300046. Epub 2023 Jul 20. PMID 38145006